CLINICAL TRIAL: NCT06006897
Title: Pain, Physical Activity, Posture and Quality of Life in Individuals With Idiopathic Scoliosis Who Have Had COVID-19
Brief Title: Pain, Physical Activity, Posture and Quality of Life in Post-COVID-19 Individuals With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Associate Professor, Principal Investigator, Izmir Democracy University
Other Study IDs: Effects of COVID on scoliosis
Record Dates: First submitted 2023-08-21; First posted 2023-08-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Respiratory Infection; Idiopathic Scoliosis
Keywords: pain; physical activity; posture; quality of life; Scoliosis
MeSH Terms: conditions — Pain; Motor Activity; Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID-19 group: This group will consist of individuals with idiopathic scoliosis who have had COVID-19.
  Interventions: Other: Physical Evaluations of post-COVID-19 individuals
- Control group: The control group will consist of individuals with idiopathic scoliosis without post-COVID-19.
  Interventions: Other: Physical evaluations of non-post-COVID-19 individuals

INTERVENTIONS:
Other: Physical Evaluations of post-COVID-19 individuals — In this study, scoliosis degree measurement, number of steps, pain, posture and quality of life will be evaluated in idiopathic scoliosis with post-COVID-19 individuals. The data to be obtained from all these evaluations will be collected from the individuals at one time and over a period of approximately 1 hour at the most. Step count tracking with pedometer will be done for each individual for 3 days.
  Groups: Post-COVID-19 group
Other: Physical evaluations of non-post-COVID-19 individuals — In this study, scoliosis degree measurement, number of steps, pain, posture and quality of life will be evaluated in idiopathic scoliosis without post-COVID-19 individuals.
  Groups: Control group

SUMMARY:
It is not known to what extent the COVID-19 virus affects individuals with scoliosis during the prolonged COVID-19 pandemic. Therefore, in this study it was aimed to comparatively investigate pain severity, posture disorders that can be assessed by artificial intelligence, physical activity levels and quality of life in individuals with idiopathic scoliosis with and without COVID-19.

DETAILED DESCRIPTION:
Various physical and psychological disorders observed in individuals with scoliosis have worsened during the pandemic period. However, it is still not fully known to what extent the COVID-19 virus affects individuals with scoliosis during the prolonged COVID-19 pandemic. For this reason, this study aimed to comparatively investigate pain severity, posture disorders that can be assessed by artificial intelligence, physical activity levels and quality of life in individuals with idiopathic scoliosis with and without COVID-19.

With the findings obtained from this way, it is expect that artificial intelligence technology will shed light on a new approach to the rehabilitation of individuals with idiopathic scoliosis who have suffered from COVID-19. In addition, if there is more pain, posture disorders, physical inactivity and quality of life disorders in individuals with scoliosis who have previously experienced COVID-19, it is also aimed to bring them to light. In this way, it will be possible to provide more specific direction to the rehabilitation of these individuals.

ELIGIBILITY:
Inclusion Criteria for individuals with idiopathic scoliosis who have experienced COVID-19:

* being 18 years of age or older
* Volunteering to participate in the study
* Having been diagnosed with idiopathic scoliosis
* Being able to walk independently
* Having been diagnosed with COVID-19 and having recovered and been discharged.

Inclusion criteria for individuals with idiopathic scoliosis who have not had COVID-19;

* being 18 years of age or older
* Volunteering to participate in the study
* Being diagnosed with idiopathic scoliosis

Exclusion criteria for individuals with idiopathic scoliosis who have had COVID-19;

* Having been diagnosed with COVID-19 in the last 15 days
* Being suspected of COVID-19
* Having mental problems that may affect cooperation
* Having an acute or chronic infection that may affect the evaluations to be made within the scope of the study.
* Participating in any professional sports activity
* Having any surgery to prevent walking, having a chronic disease, orthopedic/neurological/cardiopulmonary disease, physical or mental disability and/or cognitive impairment
* Using analgesics and other interactive drugs that will affect assessments
* Being pregnant

Exclusion criteria for individuals with idiopathic scoliosis who have not had COVID-19;

* Having had at least one COVID-19
* Being suspected of COVID-19
* Having any mental or physical disability
* Having any acute or chronic illness
* Having analgesic drug use that will affect the evaluations . Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 25 idiopathic scoliosis with post-COVID-19 will be included in the main group and at least 25 idiopathic scoliosis without post-COVID-19 will be included in control group.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Daily average step count | through study completion, an average of 1 year
  The step counts will be recorded via pedometers everyday within 3 days after confirming enrolment.

SECONDARY OUTCOMES:
Pain Intensity measured with the Numerical Rating Scale. | through study completion, an average of 1 year
  Pain intensity will be measured with the Numerical Rating Scale. This scale expresses the severity of pain with integers from 0 (no pain) to 10 (the worst possible pain).
Total quality of life score evaluated by Scoliosis Research Society-22 (SRS-22) questionnaire. | through study completion, an average of 1 year
  The score will be evaluated using Scoliosis Research Society-22 (SRS-22) questionnaire. SRS-22 contains 22 questions. Each question is scored from 1 (worst) to 5 (best), with higher scores indicating better results. The minimum score obtained from the questionnaire is 22 and the maximum total score is 110.
Posture assessment | through study completion, an average of 1 year
  Posture deviation will be determined according to the deviation score in the joint centers obtained by photographing the posture of the individuals and uploading them to the system. Posture assessment will be made with a mobile application based on the concept of postural analysis with artificial intelligence.
Degree of vertebral rotation | through study completion, an average of 1 year
  Degree of vertebral rotation will be evaluated through a scoliometer.
Pain severity | through study completion, an average of 1 year
  Pain severity will be assessed via Pressure Algometry

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Study Director — Izmir Democracy University; MERVE NUR YÜKSEL, Principal Investigator — Izmir Democracy University; ALİ ERTUĞRUL, Principal Investigator — Balikesir Ataturk City Hospital; RUKİYE YAZICI, Principal Investigator — Atatürk, Balikesir State Hospital
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kieser DC, Bourghli A, Larrieu D, Cawley DT, Hayashi K, Jakinapally S, Pizones J, Boissiere L, Obeid I. Impact of COVID-19 on the pain and disability of patients with adult spinal deformity. Spine Deform. 2021 Jul;9(4):1073-1076. doi: 10.1007/s43390-021-00315-5. Epub 2021 Mar 2. PMID 33651340
- [Background] Suarez-Huerta ML, Gomez-Rice A, Carvajal Alvarez M, Vazquez Vecilla IC, Izquierdo-Nunez E, Fernandez-Gonzalez M, Zuniga-Gomez L, Betegon-Nicolas J, Sanchez-Campos S. Effect of COVID-19 on quality of life of persons aged >70 years with adult spinal deformity: A cross-sectional case-control study. Medicine (Baltimore). 2022 Aug 19;101(33):e29954. doi: 10.1097/MD.0000000000029954. PMID 35984207